CLINICAL TRIAL: NCT03679767
Title: A Phase 2 Study of INCMGA00012 (PD-1 Inhibitor) in Participants With Selected Solid Tumors (POD1UM-203)
Brief Title: A Study of INCMGA00012 in Participants With Selected Solid Tumors (POD1UM-203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-203
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Non-small Cell Lung Cancer; Locally Advanced Urothelial Cancer; Metastatic Urothelial Cancer; Unresectable Melanoma; Metastatic Melanoma; Locally Advanced Renal Cell Carcinoma; Metastatic Clear-Cell Renal Cell Carcinoma
Keywords: PD-1inhibitor; non-small cell lung cancer; urothelial cancer; melanoma; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Melanoma: retifanlimab 500 mg (Experimental): Participants with melanoma received retifanlimab 500 milligrams (mg) every 4 weeks (Q4W), administered by intravenous (IV) infusion over 30 minutes on Day 1 of each 28-day cycle.
  Interventions: Drug: Retifanlimab
- NSCLC: retifanlimab 500 mg (Experimental): Participants with non-small cell lung cancer (NSCLC) received retifanlimab 500 mg Q4W, administered by IV infusion over 30 minutes on Day 1 of each 28-day cycle.
  Interventions: Drug: Retifanlimab
- UC: retifanlimab 500 mg (Experimental): Participants with urethelial carcinoma (UC) received retifanlimab 500 mg Q4W, administered by IV infusion over 30 minutes on Day 1 of each 28-day cycle.
  Interventions: Drug: Retifanlimab
- RCC: retifanlimab 500 mg (Experimental): Participants with renal cell carcinoma (RCC) received retifanlimab 500 mg Q4W, administered by IV infusion over 30 minutes on Day 1 of each 28-day cycle.
  Interventions: Drug: Retifanlimab

INTERVENTIONS:
Drug: Retifanlimab — Retifanlimab administered intravenously at 500 mg every 4 weeks
  Other Names: INCMGA00012

SUMMARY:
The purpose of this study is to assess the clinical activity and safety of INCMGA00012 in participants with advanced solid tumors where the efficacy of PD-1 inhibitors has previously been established.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following: treatment-naïve metastatic non-small cell lung cancer with high PD-L1 expression (tumor proportion score ≥ 50%) and no epidermal growth factor receptor (EGFR), alkaline phosphatase (ALK), or ROS activating genomic tumor aberrations; locally advanced or metastatic urothelial carcinoma in participants who are not eligible for cisplatin therapy and whose tumors express PD-L1 with a combined positive score ≥ 10; unresectable or metastatic melanoma; locally advanced or metastatic renal cell carcinoma with clear cell component (with or without sarcomatoid features) and having received no prior systemic therapy.
* Measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Receipt of anticancer therapy or participation in another interventional clinical study within 21 days before the first administration of study drug.
* Prior treatment with PD-1 or PD-L1 directed therapy (other immunotherapies may be acceptable with prior approval from the medical monitor).
* Radiotherapy within 14 days of first dose of study treatment with the following caveats: 28 days for pelvic radiotherapy; 6 months for thoracic region radiotherapy that is > 30 Gy.
* Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of anemia not requiring transfusion support and any grade of alopecia). Endocrinopathy, if well-managed, is not exclusionary and should be discussed with sponsor medical monitor.
* Has not recovered adequately from toxicities and/or complications from surgical intervention before starting study drug.
* Laboratory values outside the protocol-defined range at screening.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 3 years of study entry.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg of prednisone or equivalent).
* Evidence of interstitial lung disease or active noninfectious pneumonitis.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Known active hepatitis B antigen, hepatitis B virus, or hepatitis C virus infection.
* Active infections requiring systemic therapy.
* Known to be HIV-positive, unless all of the following criteria are met: CD4+ count ≥ 300/μL, undetectable viral load, receiving antiretroviral therapy.
* Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Impaired cardiac function or clinically significant cardiac disease.
* Is pregnant or breastfeeding.
* Has received a live vaccine within 28 days of the planned start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cornfeld, MD, Study Director — Incyte Corporation
Locations (52):
- United States (18):
  - California Cancer Associates for Research and Excellence, Inc., Fresno, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - California Cancer Associates for Research and Excellence, Inc., San Marcos, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - St. Joseph Health Medical Group - Annadel Medical Group, Santa Rosa, California
  - Rocky Mountain Cancer Centers - Denver - Midtown, Denver, Colorado
  - Christiana Care Helen F. Graham Cancer Center, Newark, Delaware
  - Rcca Md, Llc, Bethesda, Maryland
  - VA New Jersey Health Care System, East Orange, New Jersey
  - New York Oncology Hematology - Albany, Albany, New York
  - Kaiser Permanente, Portland, Oregon
  - Texas Oncology Surgical Specialists - Austin Central, Austin, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - AIM Trials, LLC, Plano, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., The Woodlands, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Wytheville, Virginia
- Austria (4):
  - LKH Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Ordensklinikum, Linz
  - Universitatsklinikum St. Polten, Sankt Pölten
- France (5):
  - Institut Bergonié, Bordeaux
  - Institut Paoli Calmettes, Marseille
  - CEPCM / CHU Timone, Marseille
  - Georges Pompidou European Hospital, Paris
  - Hopitaux Universitaires De Strasbourg, Strasbourg
- Hungary (2):
  - BAZ County Hospital, Miskolc
  - Hetenyi G Korhaz, Onkologiai Kozpont, Szolnok
- Italy (5):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti di Ancona, Ancona
  - ASST Istituti Ospitalieri, Cremona
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
- Poland (4):
  - Med-Polonia Sp. z o. o., Poznan, Greater Poland Voivodeship
  - Centrum Onkologii- Instytut im Marii Skłodowskiej Curie, Warsaw, Masovian Voivodeship
  - Specjalistyczna Praktyka Lekarska, Lublin
  - BioVirtus Research Site, Otwock
- Romania (7):
  - Centrul de Oncologie Sfantul Nectarie, Craiova, Dolj
  - Oncolab SRL, Craiova, Dolj
  - Medisprof SRL, Cluj-Napoca
  - Clinical Emergency Hospital of Constanta, Constanța
  - Center of Oncology Euroclinic, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Oncocenter - Oncologie Clinica SRL, Timișoara
- Spain (7):
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Centro Oncologico De Galicia, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Puerta De Hierro, Majadahonda
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 study centers in Austria, Spain, France, Hungary, Italy, Poland, Romania, and the United States.
Pre-assignment Details: A total of 121 participants with advanced solid tumors (melanoma, non-small cell lung cancer, urethelial carcinoma, and renal cell carcinoma) were enrolled in the study and treated with retifanlimab.
Groups:
- Melanoma: Participants with melanoma received retifanlimab 500 milligrams (mg), administered by intravenous (IV) infusion over 30 minutes on Day 1 of each 28-day cycle (Q4W).
- Non-small Cell Lung Cancer: Participants with non-small cell lung cancer received retifanlimab 500 mg, administered by IV infusion over 30 minutes on Day 1 Q4W.
- Urethelial Carcinoma: Participants with urethelial carcinoma received retifanlimab 500 mg, administered by IV infusion over 30 minutes on Day 1 Q4W.
- Renal Cell Carcinoma: Participants with renal cell carcinoma received retifanlimab 500 mg, administered by IV infusion over 30 minutes on Day 1 Q4W.
Period: Overall Study
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Started | 35 | 23 | 29 | 34
Completed | 0 | 0 | 0 | 0
Not Completed | 35 | 23 | 29 | 34
Not completed — Death | 16 | 11 | 17 | 10
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Follow-up Completed | 18 | 11 | 11 | 20
Not completed — Entered Hospice Care | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma | Total
Number analyzed (Participants) | 35 | 23 | 29 | 34 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (15.24) | 67.8 (8.68) | 72.0 (8.23) | 66.6 (10.28) | 68.3 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 7 | 4 | 10 | 41
  Male | 15 | 16 | 25 | 24 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 35 | 22 | 20 | 33 | 110
  Asian | 0 | 1 | 0 | 0 | 1
  Not Reported | 0 | 0 | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 30 | 22 | 12 | 29 | 93
  Not Reported | 1 | 1 | 16 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1), as determined by the investigator, at any post-Baseline visit until new anti-cancer therapy or first Progressive Disease. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 25.9 months
Population: Full Analysis Set (FAS) Population: all study participants who had received at least 1 dose of study drug. Participants were to be analyzed based on disease-specific diagnosis. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 35 | 23 | 29 | 34
percentage of participants | 40.0 [23.9 to 57.9] | 34.8 [16.4 to 57.3] | 37.9 [20.7 to 57.7] | 23.5 [10.7 to 41.2]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from initial objective response (CR or PR) per RECIST v1.1 until the first observation of documented disease progression (PD), as determined by the investigator, or death due to any cause. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 24.0 months
Population: FAS Population. Only those participants with a CR or PR were included in the analysis. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 14 | 8 | 11 | 8
months | NA [9.2 to NA] — The median and upper limit of the confidence interval were not estimable because too few participants had events of disease progression or death. | 18.2 [1.9 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of disease progression or death. | 11.5 [2.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of disease progression or death. | NA [2.8 to NA] — The median and upper limit of the confidence interval were not estimable because too few participants had events of disease progression or death

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with an overall response of CR, PR, or stable disease (SD), per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 25.9 months
Population: FAS Population. Confidence intervals were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 35 | 23 | 29 | 34
percentage of participants | 54.3 [36.6 to 71.2] | 65.2 [42.7 to 83.6] | 55.2 [35.7 to 73.6] | 64.7 [46.5 to 80.3]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: According to RECIST 1.1, PFS was defined as the length of time from the initial infusion of study drug until the earliest date of disease progression, determined by investigator assessment, or death due to any cause, if occurring sooner than progression.
Time Frame: up to 25.9 months
Population: FAS Population. Median PFS was estimated using the Kaplan-Meier method. The confidence interval for median PFS was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 35 | 23 | 29 | 34
months | 3.6 [1.8 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of disease progression or death. | 4.4 [1.8 to 21.9] | 5.7 [1.8 to 13.6] | 5.4 [2.3 to 11.4]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months between the first dose date (Day 1) and the date of death due to any cause.
Time Frame: up to 28.2 months
Population: FAS Population. Median survival time in months was estimated using the Kaplan-Meier method. The confidence interval for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 35 | 23 | 29 | 34
months | NA [8.7 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had events of death. | 21.9 [5.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of death. | 15.2 [7.7 to NA] — The upper limit of the confidence interval was not estimable because too few participants had events of death. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had events of death.

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of retifanlimab and until the earlier of 90 days of the last administration of retifanlimab and new anti-cancer therapy start if any, are reported.
Time Frame: up to approximately 2.3 years
Population: Safety Evaluable Population: all participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urethelial Carcinoma | Renal Cell Carcinoma
Number analyzed (Participants) | 35 | 23 | 29 | 34
Participants | 32 | 21 | 28 | 32

7. Secondary Outcome: First-dose Cmax of Retifanlimab
Description: Cmax was defined as the maximum observed plasma or serum concentration of retifanlimab.
Time Frame: preinfusion and 10 minutes postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of study drug and provided a Baseline and at least 1 postdose PK sample
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Groups:
- All Participants: Participants with melanoma, non-small cell lung cancer, urethelial carcinoma, and renal cell carcinoma received retifanlimab 500 mg, administered by IV infusion over 30 minutes on Day 1 Q4W.
Arm/Group | All Participants
Number analyzed (Participants) | 121
milligrams per Liter (mg/L) | 143 (30.9)

8. Secondary Outcome: Cmax of Retifanlimab at Steady-state
Description: Cmax was defined as the maximum observed plasma or serum concentration of retifanlimab.
Time Frame: preinfusion and 10 minutes postinfusion (± 10 minutes) on Day 1 of Cycles 1, 2, 4, and 6 (up to approximately 168 days; each cycle was 28 days)
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 121
mg/L | 181 (39.4)

9. Secondary Outcome: First-dose Tmax of Retifanlimab
Description: tmax was defined as the time to the maximum concentration of retifanlimab.
Time Frame: preinfusion and 10 minutes postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: PK Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 121
hours | 0.500 [0.500 to 1.00]

10. Secondary Outcome: Tmax of Retifanlimab at Steady-state
Description: tmax was defined as the time to the maximum concentration of retifanlimab.
Time Frame: as for outcome 8
Population: PK Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 121
hours | 0.500 [0.500 to 1.00]

11. Secondary Outcome: First-dose Cmin of Retifanlimab
Description: Cmin was defined as the minimum observed plasma or serum concentration over the dose interval of retifanlimab.
Time Frame: preinfusion and 10 minutes postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 121
mg/L | 18.0 (7.52)

12. Secondary Outcome: Cmin of Retifanlimabv at Steady-state
Description: Cmin was defined as the minimum observed plasma or serum concentration over the dose interval of retifanlimab.
Time Frame: as for outcome 8
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 121
mg/L | 38.2 (16.3)

13. Secondary Outcome: First-dose AUC0-t of Retifanlimab
Description: AUC0-t was defined as the area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t of retifanlimab.
Time Frame: preinfusion and 10 minutes postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: day*mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 121
day*mg/L | 1620 (506)

14. Secondary Outcome: AUC0-t of Retifanlimab at Steady-state
Description: as for outcome 13
Time Frame: as for outcome 8
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: day*mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 121
day*mg/L | 2030 (566)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for up to approximately 2.3 years. All-Cause Mortality was assessed for up to 28.2 months
Description: Treatment-emergent adverse events, defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of retifanlimab and until the earlier of 90 days of the last administration of retifanlimab and new anti-cancer therapy start if any, are reported.
Groups:
- Urothelial Cancer: Participants with urethelial carcinoma received retifanlimab 500 mg, administered by IV infusion over 30 minutes on Day 1 Q4W.
- Total: Total
Arm/Group | Melanoma | Non-small Cell Lung Cancer | Urothelial Cancer | Renal Cell Carcinoma | Total
All-Cause Mortality (participants affected / at risk) | 16/35 | 11/23 | 17/29 | 10/34 | 54/121
Serious Adverse Events (participants affected / at risk) | 8/35 | 9/23 | 12/29 | 11/34 | 40/121
Other Adverse Events (participants affected / at risk) | 30/35 | 19/23 | 25/29 | 30/34 | 104/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma (N=35) | Non-small Cell Lung Cancer (N=23) | Urothelial Cancer (N=29) | Renal Cell Carcinoma (N=34) | Total (N=121)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melanoma (N=35) | Non-small Cell Lung Cancer (N=23) | Urothelial Cancer (N=29) | Renal Cell Carcinoma (N=34) | Total (N=121)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 7 (8)
Amylase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 9 (9) | 5 (5) | 17 (17)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 0 (0) | 8 (15) | 5 (13) | 21 (38)
Asthenia (General disorders) | 7 (11) | 2 (2) | 9 (11) | 6 (7) | 24 (31)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (3) | 10 (11)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 2 (3) | 9 (10)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (9) | 5 (5) | 14 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 1 (4) | 4 (4) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 7 (8) | 3 (3) | 19 (20)
Diarrhoea (Gastrointestinal disorders) | 7 (22) | 3 (3) | 5 (6) | 4 (7) | 19 (38)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (3) | 4 (5) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (3) | 1 (1) | 6 (6) | 12 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (4) | 5 (8)
Fatigue (General disorders) | 6 (7) | 2 (2) | 2 (2) | 2 (2) | 12 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 1 (2) | 1 (1) | 0 (0) | 9 (10)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 5 (6)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 3 (4) | 2 (2) | 6 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Hypothyroidism (Endocrine disorders) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 11 (11)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Malaise (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 4 (4) | 3 (3) | 12 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (4)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (4) | 10 (11)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 2 (2) | 8 (10)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 8 (8)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 4 (6) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12) | 3 (3) | 4 (5) | 5 (5) | 21 (25)
Pyrexia (General disorders) | 3 (6) | 2 (2) | 4 (7) | 4 (8) | 13 (23)
Rash (Skin and subcutaneous tissue disorders) | 5 (12) | 2 (2) | 3 (3) | 5 (5) | 15 (22)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 3 (5)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 5 (6) | 4 (5) | 5 (6) | 17 (21)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vitiligo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (4) | 1 (1) | 6 (9)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT03679767/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT03679767/SAP_001.pdf